CLINICAL TRIAL: NCT03058939
Title: Assessing the REsponse Rate of Weekly Neo-adjuvanT pacliTAxel (Taxol) in Nigerian Women With Breast Cancer (ARETTA)
Brief Title: Assessing the Response Rate of Neo-adjuvant Paclitaxel (Taxol) in Nigerian Women With Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never activated to enrollment.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1005
Record Dates: First submitted 2017-02-02; First posted 2017-02-23 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III; Paclitaxel; Taxol
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; pertuzumab; Trastuzumab; Tamoxifen; Letrozole; Gonadotropin-Releasing Hormone; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Paclitaxel (Experimental): Investigators plan to treat patients with paclitaxel weekly for a total of approximately 16 weeks (8 weeks before ultrasonography for response assessment and 8 weeks before surgery in good responders). Paclitaxel 80mg/m2 will be given on days 1, 8, 15 and so on for a total of 8 doses.
  Interventions: Drug: Paclitaxel
- Carboplatin (Other): After first 8 weeks of paclitaxel, those with progressive disease (based on breast US assessment) or partial response but inoperable will have carboplatin added to their regimen. Patients will receive 8 cycles of weekly paclitaxel and carboplatin (PC).
  Interventions: Drug: Carboplatin
- Fluorouracil Epirubicin Hydrochloride Cyclophonsphamide (FEC) (Other): Patients with poor response to 8 courses of paclitaxel followed by 8 courses of PC based on ultrasound assessment will be regarded as failing to respond to treatment. These patients will receive 4 cycles of 3-weekly FEC and will be followed up.
  Interventions: Drug: FEC
- LHRH (luteinizing hormone-releasing hormone) (Other): All Premenopausal patients will receive LHRH agonist for two years for contraception and fertility preservation.
  Interventions: Drug: LHRH agonist
- Tamoxifen or letrozole (Other): Hormone-receptor positive patients will receive hormonal therapy with tamoxifen or letrozole after surgery, radiotherapy and LHRH agonist according to the expression of hormone receptors and according to the state of primary menopause at the onset of the study.
  Interventions: Drug: Tamoxifen; Drug: Letrozole
- Herceptin SC and Perjeta (Other): Patients with HER2-positive disease (see glossary and section 10.3) will receive 5 three-weekly courses of trastuzumab (Herceptin SC) with pertuzumab (Perjeta). After that pts will continue receiving trastuzumab to complete total of 18 doses within 1 year of treatment.
  Interventions: Drug: Perjeta; Drug: Herceptin SC

INTERVENTIONS:
Drug: Paclitaxel — Administered to all patients for a minimum of 8 doses with a possible maximum of 16 doses.
  Other Names: Taxol
  Arms: Paclitaxel
Drug: Perjeta — Only administered to patients with HER2-positive disease.
  Other Names: Pertuzumab
  Arms: Herceptin SC and Perjeta
Drug: Herceptin SC — Only administered to patients with HER2-positive disease.
  Other Names: Trastuzumab
  Arms: Herceptin SC and Perjeta
Drug: Tamoxifen — Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
  Arms: Tamoxifen or letrozole
Drug: Letrozole — Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
  Arms: Tamoxifen or letrozole
Drug: LHRH agonist — Administered to all premenopausal patients.
  Arms: LHRH (luteinizing hormone-releasing hormone)
Drug: FEC — Only administered to patients who received paclitaxel and carboplatin, and were assessed as having poor response (defined as stable disease or progressive disease or partial response inoperable).
  Arms: Fluorouracil Epirubicin Hydrochloride Cyclophonsphamide (FEC)
Drug: Carboplatin — Only administered to patients who receive paclitaxel and were assessed as having poor response (defined as stable disease or progressive disease or partial response inoperable).
  Arms: Carboplatin

SUMMARY:
This is a two-stage phase II study with a single arm design. It will be conducted in women with breast cancer with stages IIA to IIIC (defined by AJCC 2009 classification) of all histological subtypes. All patients will receive 16 doses of paclitaxel; three breast ultrasound tests and tumor pathologic response evaluation will be used to assess the response to treatment.

DETAILED DESCRIPTION:
Each patient will be assigned one of the following groups: 1) complete response, 2) partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 8) unknown (not assessable, insufficient data). Patients with a good response to 8 doses of paclitaxel (complete response or partial response that are operable) will receive an additional 8 courses of paclitaxel chemotherapy before surgery and radiotherapy. The overall response for these patients will be assessed by ultrasonography after a total of 16 weeks of Taxol therapy. Patients with poor response (defined as stable disease or progressive disease or partial response inoperable) as best response after eight weekly courses of paclitaxel will receive 8 cycles of weekly PC. The overall response for these patients will also be assessed by ultrasonography after 8 courses of PC therapy. Patients with poor response to 8 courses of paclitaxel followed by 8 courses of PC based on ultrasound assessment will be regarded as failing to respond to treatment. These patients will receive 4 cycles of 3-weekly FEC and will be followed up. Patients in response groups 4-8 above will be considered as failing to respond to treatment.

All conclusions will be based on all eligible patients. The schema for the study is presented in Figures 4-1, 4-2 and 4-3. Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time will be classified as having "symptomatic deterioration". Every effort will be made to document the objective progression even after discontinuation of treatment. All Premenopausal patients will receive LHRH agonist for two years for contraception and fertility preservation. Hormone-receptor positive patients will receive hormonal therapy with tamoxifen or letrozole after surgery, radiotherapy and LHRH agonist according to the expression of hormone receptors ER and PgR (see glossary and section 10.3) and according to the state of primary menopause (see glossary) at the onset of the study. Patients with HER2-positive disease (see glossary and section 10.3) will receive 5 threeweekly courses of trastuzumab (Herceptin SC) with pertuzumab (Perjeta). After that pts will continue receiving trastuzumab to complete total of 18 doses within 1 year of treatment.

The study is designed to estimate the RR of breast cancer patients to weekly paclitaxel chemotherapy and to determine the RR to weekly PC combination chemotherapy in patients resistant to or with poor response (including early progression) while on weekly single agent paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages of 18 to 70 years old.
2. Biopsy-accessible breast tumor of significant size for core needle biopsy (≥ 2cm).
3. Patients with histologically confirmed carcinoma of the female breast with any or unknown HRs/HER2 status
4. Clinical stages IIA -IIIC. (AJCC 2009) (Appendix A)
5. Chemotherapy-naïve patients (for this malignancy)
6. Performance status: ECOG performance status 0-3 (Appendix B)
7. Non-pregnant and not nursing. Women of childbearing potential must take the pregnancy test and must commit to receive LHRH agonist Zoladex (goserelin) for two years starting from the commencement of the study medications.
8. Required Initial Laboratory Data. Adequate hematologic, renal and hepatic function, as defined by each of the following:

   1. Granulocyte ≥ 1,500/μL
   2. Platelet count ≥ 100,000/μL
   3. Absolute neutrophil count (ANC) ≥ l500/μL
   4. Hemoglobin³10g/dL
   5. Bilirubin ≤ 1.5 x upper limit of normal
   6. SGOT and SGPT < 2.5 x upper limit of normal for patients without liver metastases
   7. Creatinine within institutional normal limits or glomerular filtration rate ≥ 30 mL/min/1.73 m2 by CKD EPI equation (see http://mdrd.com/ for calculator)

Exclusion Criteria:

1. Pregnant or lactating women. Women of childbearing potential not using a reliable and appropriate contraceptive method. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.

   Patients will agree to continue the use of acceptable form of contraception for 30 days from the date of last drug administration.
2. Patients with brain metastasis.
3. Serious, uncontrolled, concurrent infection(s).
4. Patients who have received more than 4 weeks of tamoxifen therapy for this malignancy. Patient who have received tamoxifen or raloxifene for purposes of chemoprevention (e.g. Breast Cancer Prevention Trial or for other past indications (including previous breast cancer) are eligible. Tamoxifen or raloxifene therapy will be discontinued at least one month before the patient is enrolled on this study.
5. Treatment for other carcinomas within the last 5 years, except non-melanoma skin cancer and treated cervical carcinoma in-situ (CCIS).
6. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
7. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation including but not limited to chronic or active infection, HIV-positive patient, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled Diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Unwillingness to participate or inability to comply with the protocol for the duration of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Measure overall clinical response rate (OCR) | 24 months
  OCR will be calculated as the proportion of patients with an overall response of complete clinical response (CCR) or partial clinical response (PCR), where tumor response is based on change in tumor diameter after treatment.
Measure of complete pathologic response (pCR) | 24 months
  The absence of residual invasive disease in the breast and in the axillary lymph nodes at the completion of treatment will be measured.

SECONDARY OUTCOMES:
Number of participants with adverse events | 24 months
  Incidence and severity of adverse drug reactions (AE) and serious adverse drug reactions (SAE) including clinical laboratory values, vital signs, ECGs and dose interruptions.
Time until progression free survival (PFS) | From start date of therapy to the date of first documented disease progression or death from any cause, whichever may come first, assessed up to 100 months
Duration of response (DOR) | From first reponse to the date of first documented disease progression, assessed up to 24 months
Analysis of changes from baseline using the quality of life (QoL) instrument | From start date of therapy to the date of first documented disease progression or death from any cause, whichever may come first, assessed up to 100 months.
  The various domains of QoL over time and the changes from baseline using the validated (by the European Organization for Research and Treatment of Cancer (EORTC)) QoL instrument (global and breast module).
To assess the genetic and epigenetic factors associated with breast cancer in Nigeria | From start date of therapy to the date of death from any cause, assessed up to 100 months
  Through correlative study of molecular markers and tumor subtypes/tumor biology with patient's characteristics, response to treatment and patients' outcome
Blood concentrations of Perjeta before each dose of Perjeta/Herceptin/paclitaxel/PC | 24 months
  To determine the profile of Perjeta given in combination with Herceptin SC, paclitaxel and paclitaxel + carboplatinum
Blood concentrations of Herceptin SC before each dose of Herceptin/paclitaxel/PC | 24 months
  To determine the profile of Herceptin SC given in combination with Perjeta, paclitaxel and PC
Analysis of hormone recepters (ER and PgR) and HER2 | Through study completion an average of two years
  To determine the pattern of response to weekly paclitaxel and PC in combination with hormone therapy or with H/Ptz dual anti-HER2 blockade based on status of clinical markers ! Hormone receptors (ER and PgR) and HER2, and other markers.

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo I. Olopade, MD, Principal Investigator — University of Chicago Center for Global Health
Locations (1):
- Lagos State University College of Medicine, Ikeja, Lagos, Nigeria